CLINICAL TRIAL: NCT03441100
Title: Phase 1 Study Evaluating Genetically Modified Autologous T Cells Expressing a T-cell Receptor Recognizing a Cancer/Germline Antigen in Patients With Recurrent and/or Refractory Solid Tumors(ACTengine® IMA202-101)
Brief Title: TCR-engineered T Cells in Solid Tumors: IMA202-101
Acronym: ACTengine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immatics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMA202-101
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor, Adult; Refractory Cancer; Recurrent Cancer; Cancer
Keywords: T-Cell therapy; Immunotherapy; Adoptive cellular therapy; T-Cell Receptor; Cell Therapy; Cytotherapy; IMA202
MeSH Terms: conditions — Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental: IMA202 Product (Experimental): * Pre-conditioning by non-myeloablative chemotherapy with Fludarabine and Cyclophosphamide
  * One dose of IMA202 product will be infused intravenously. Four dose levels will be evaluated. At least two patients per cohort will be treated.
  * Post-infusion of IMA202 product, administration of low dose recombinant human interleukin-2
  Interventions: Drug: IMA202 Product; Device: IMADetect®

INTERVENTIONS:
Drug: IMA202 Product — The cell dose will be based on viable CD3+CD8+ HLA-Dextramer+ cells per body surface area (BSA) as defined by the Mosteller formula.
Device: IMADetect® — IMADetect® is developed as a companion diagnostic to aid in selecting patients with relapsed and/or refractory solid cancers who might be eligible for enrollment in clinical trials. IMADetect® is intended for investigational use only.

SUMMARY:
The study purpose is to establish the safety and tolerability of IMA202 product in patients with solid tumors that express melanoma-associated antigen 1 (MAGEA1).

DETAILED DESCRIPTION:
SCREENING: Patient eligibility will be determined by HLA (human leukocyte antigen) screening and a biopsy for biomarker screening. If the patient is eligible, white blood cells will be taken during leukapheresis for the manufacture of the IMA202 product.

MANUFACTURING: IMA202 product will be made from the patient's white blood cells.

TREATMENT: Lymphodepletion with cyclophosphamide and fludarabine will occur in the days before the IMA202 product infusion to improve the duration of time that IMA202 product stays in the body. The patient will be admitted to the hospital during the treatment.

After the IMA202 product infusion, a low dose of IL-2 will be given twice daily for a period of time.

Patients will be closely monitored for safety and for a total of 3 years post IMA202 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced and/or metastatic solid tumor
* Patients may enter screening procedure before, during, or after the last available indicated standard of care treatment. There is no limitation for prior anti cancer treatments.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* HLA phenotype positive for the study
* Measurable disease and accessible to biopsy
* Adequate pulmonary function per protocol
* Acceptable organ and bone marrow function per protocol
* Acceptable coagulation status per protocol
* Adequate hepatic function per protocol
* Adequate renal function per protocol
* Patient's tumor must express tumor antigen by qPCR using a fresh tumor biopsy specimen
* Life expectancy more than 3 months
* Confirmed availability of production capacities for IMA202 product
* Patients must have recurrent/progressing and/or refractory solid tumors and must have received or not be eligible for all available indicated standard of care treatment.
* For hepatocellular carcinoma (HCC) patients only, Child-Pugh score of ≤ 6
* IMA202 product must have passed all of the release tests
* Female patient of childbearing potential must use adequate contraception prior to study entry until 12 months after the infusion of IMA202
* Male patient must agree to use effective contraception or be abstinent while on study and for 6 months after the infusion of IMA202
* Hepatocellular carcinoma (HCC) patients with liver cirrhosis only - upper endoscopy is required within 6 months of study entry
* The patient must have recovered from any side effects of prior therapy to Grade 1 or lower (except for non-clinically significant toxicities; e.g., alopecia, vitiligo) prior to lymphodepletion. As determined by the investigator, the patient may still be eligible if the patient has not fully recovered from Grade ≥ 2 toxicities if these toxicities are not anticipated to further improve (e.g., chronic neuropathy) and such toxicities are not anticipated to worsen with the lymphodepletion therapy

Exclusion Criteria:

* History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years
* Solid tumors with low likelihood of tumor biomarker expression per protocol
* Pregnant or breastfeeding
* Serious autoimmune disease Note: At the discretion of the investigator, these patients may be included if their disease is well controlled without the use of immunosuppressive agents.
* History of cardiac conditions as per protocol
* Prior stem cell transplantation or solid organ transplantation
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study
* History of hypersensitivity to cyclophosphamide (CY), fludarabine (FLU), IL-2, or any of the rescue medications
* History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician
* HIV infection, active hepatitis B virus (HBV), active hepatitis C virus (HCV) infection, ongoing active anti-HCV treatment or detectable HBV or HCV viral load at the most recent laboratory report. Patients with both HBV and HCV infections will be excluded from screening

  1. Patients with a history of HCV infection and with an undetectable viral load per the most recent laboratory report and/or completed anti-HCV treatment but are HCV antibody positive are permitted.
  2. History of treated HBV infection is permitted if the viral load is undetectable per the most recent laboratory report. Note: HCC patients with controlled HBV infection, as defined by resolved (anti-hepatitis B surface antigen [HBs-Ag] antibody (Ab) negative, anti-core antigen [HBc Ag] Ab positive) or chronic stable (anti HBs-Ag Ab positive) HBV infection will be eligible for screening. Patients with active HBV infection who are not on anti-HBV treatment will be excluded.
* Any condition contraindicating leukapheresis, lymphodepletion, low-dose IL-2, and/or IMA202 treatment
* Patients with any active viral infection
* Patients with active brain metastases

NOTE: Patients with a history of brain metastases may be eligible, if an imaging scan with contrast enhancement not older than 4 weeks is able to exclude the existence of currently active brain metastasis, and steroid therapy has been discontinued for ≥2 weeks.

* Treatment with protocol-defined excluded treatments, medical devices, and/or procedures per protocol
* Concurrent participation in an interventional part of another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | up to 3 years post treatment

SECONDARY OUTCOMES:
Persistence of T-cells | up to 3 years post treatment
Tumor response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 and immune-related RECIST (irRECIST) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cedrik Britten, MD, Study Director — Immatics US, Inc.
Locations (6):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (4):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Bonn - Medizinische Klinik III, Bonn, North Rhine-Westphalia
  - Universitätsklinikum C.-G.-Carus Dresden, Dresden, Saxony
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No